CLINICAL TRIAL: NCT00778323
Title: Effects of Remote Ischemic Preconditioning on Biochemical Markers and Neurological Outcomes in Patients Undergoing Elective Cervical Decompression Surgery
Brief Title: Clinical Trial of Remote Preconditioning in Patients Undergoing Cervical Decompression Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Lize Xiong, Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJ20070901
Record Dates: First submitted 2008-08-09; First posted 2008-10-23 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2008-11

CONDITIONS: Cervical Compression Myelopathy; Ischemia; Reperfusion Injury; Spinal Cord Injury
Keywords: remote ischemic preconditioning; cervical compression myelopathy; spinal cord; neuron-specific enolase; s-100B
MeSH Terms: conditions — Ischemia; Reperfusion Injury; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A,2, II (Experimental)
  Interventions: Procedure: limb remote ischemic preconditioning (LRIPC)

INTERVENTIONS:
Procedure: limb remote ischemic preconditioning (LRIPC) — LRIPC consists of three 5-min cycles of right upper limb ischemia induced by an automated cuff-inflator placed on the upper arm and inflated to 200 mmHg,with an intervening 5 min reperfusion during which the cuff is deflated.
  Other Names: an automated cuff-inflator made in China

SUMMARY:
The purpose of this study is to assess whether a large clinical trial testing the effect of RIPC on neurologic outcome in patients undergoing elective cervical decompression surge is warranted.

DETAILED DESCRIPTION:
Spinal cord ischemia-reperfusion injury commonly contribute to perioperative morbidity and mortality after elective cervical decompression surgery.Remote ischemic preconditioning(RIPC)is a phenomenon whereby brief periods of ischemia followed by reperfusion in one organ provide system protection from prolonged ischemia.The hypothesis of this protocol is that limb ischemic preconditioning could reduces spinal cord ischemia-reperfusion injury induced by elective cervical decompression surgery.Serum s-100B and NSE concentration will be measured before and after induction ,and at 6 hours,1,3,5 and 7days after surgery.JOA scores in all the cases will be evaluated before operation and at 7days ,1,3,6 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and radiological signs of cervical compression myelopathy(ccm)
* Age 30-75
* Stage 1-2

Exclusion Criteria:

* Age>75
* History of heart,hepatic,renal or pulmonary disease.
* History of peripheral vascular disease affecting the upper limbs.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
serum concentrations of s-100B,NSE | 1 week or more

SECONDARY OUTCOMES:
a Japanese Orthopaedic Association (JOA) scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, MD, Study Chair — Xiling Hospital,Fourth Military Medical University
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Hu S, Dong HL, Li YZ, Luo ZJ, Sun L, Yang QZ, Yang LF, Xiong L. Effects of remote ischemic preconditioning on biochemical markers and neurologic outcomes in patients undergoing elective cervical decompression surgery: a prospective randomized controlled trial. J Neurosurg Anesthesiol. 2010 Jan;22(1):46-52. doi: 10.1097/ANA.0b013e3181c572bd. PMID 19996767